CLINICAL TRIAL: NCT07222046
Title: Identifying Residual Connectivity in Veterans With Spinal Cord Injury for Precision Neurorehabilitation
Brief Title: Spinal Neurorehabilitation for Veterans With SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RRD8-003-24W
Record Dates: First submitted 2025-10-15; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal neuromodulation; Transcutaneous stimulation; Spinal cord stimulation; Neuroanatomy; Neurorehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: All participants will be Veterans with spinal cord injury to evaluate neurophysiological and functional effects of non-invasive spinal neuromodulation.
Masking Description: Due to the uniqueness of each injury, all staff will be aware of each participant's history. All participants will receive the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-arm (Experimental): This is a single-arm study where all participants will undergo the same neurophysiological, imaging, and functional testing.
  Interventions: Diagnostic Test: Neurophysiological and anatomical testing; Device: Transcutaneous Spinal Stimulation

INTERVENTIONS:
Diagnostic Test: Neurophysiological and anatomical testing — All participants will undergo neurophysiological testing (transcranial magnetic stimulation and somatosensory evoked potentials) to determine residual neural connectivity. All participants will also undergo MRI of the spine to evaluate residual neural connections and changes above and below lesion. These values will be compared to the standard clinical evaluation of spinal cord injury (ISNCSCI exam).
Device: Transcutaneous Spinal Stimulation — All participants will undergo spinal neuromodulation through non-invasive transcutaneous spinal stimulation to determine the effects on voluntary motor function, sensation, and activities of daily living.
  Other Names: Digitimer DS7

SUMMARY:
Chronic spinal cord injury (SCI) is a debilitating disorder in Veterans and the broader U.S. population that does not have a cure. Veterans with severe SCI demonstrate permanent loss of sensory and motor function below their injury resulting in decreased quality of life and independence. Recently, electrical spinal neuromodulation has emerged as a potential approach to restore voluntary motor function and locomotion in persons with chronic SCI. However, spinal neuromodulation has yet to translate to clinical use due to small sample sizes in research studies and a lack of information on which patients would benefit. Here, the investigators propose a novel approach to evaluate the priorities and barriers faced by Veterans with SCI to use spinal neuromodulation, understand the neural connections remaining in Veterans with severe SCI, and determine potential functional improvements using non-invasive spinal neuromodulation technology. This research represents the first step towards deploying techniques that could dramatically improve function and quality of life for Veterans with SCI.

DETAILED DESCRIPTION:
The International Standards for Neurological Classification of SCI (ISNCSCI) exam is used to classify spinal cord injury (SCI) severity by determining the neurological injury level and functional completeness of SCI. However, anatomical, physiological, and functional studies have indicated that many participants with ISNCSCI-defined complete SCI retain connectivity through the SCI lesion. Due to the heterogeneity of SCI and the small-N in prior spinal neuromodulation studies, there are no diagnostic criteria to determine how SCI lesion profile affects the ability to restore sensorimotor function in the presence of spinal neuromodulation. Development of this knowledge is necessary to design precise spinal neuromodulation approaches and clinical trials that could restore function and improve quality of life for Veterans with chronic SCI. First, stakeholders will be engaged to define research priorities, meaningful outcomes, and barriers to participation in neuromodulation trials. The potential impact of neuromodulation and priorities of Veterans with SCI and their caretakers will be assessed across a nationwide survey. Spinal neuromodulation will be evaluated to determine how it could impact clinical practice and treatment of Veterans though survey of SCI physicians. Qualitative feedback will be obtained from Veterans with SCI regarding the expected and achieved outcomes with neuromodulation prior to and after undergoing functional neuromodulation experiments. Next, baseline anatomical and physiological connectivity measurements across ISNCSCI scores will be established. Veterans with SCI across INSCSCI grades will be recruited to determine residual spinal connectivity. Spinal cord anatomy will be assessed above, below, and at the SCI lesion through MR neuroimaging. Descending corticospinal connectivity will be evaluated with transcranial magnetic stimulation and ascending afferent signals will be evaluated through somatosensory evoked potentials. Finally, functional spinal connectivity during spinal neuromodulation will be evaluated. Volitional motor output will be assessed with and without non-invasive spinal neuromodulation. The sensory effects of spinal neuromodulation will be assessed through user reports of pain and somatosensation. Potential functional improvements in activities of daily living will be assessed with and without spinal neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be able to independently read and understand study information materials necessary to ensure informed consent.
* All participants must have a chronic spinal cord injury occurring >1 year prior to study enrollment.
* Ability to follow simple commands in English.

Exclusion Criteria:

* Contraindications to the use of external magnetic or electrical stimulation (e.g., epilepsy, intracranial metal, implanted electrosensitive device, etc.)
* Significant neurological comorbidities that may affect neurophysiological recordings
* Functional disability prior to spinal cord injury
* Visual or auditory disorders limiting ability to participate in study procedures
* Pregnancy
* Primary psychiatric disorders or dissociative mental symptoms that impair informed consent
* Significant chronic pain that may preclude an MRI scan or performing neurorehabilitation exercises
* Frequent and significant spasticity that may preclude an MRI scan or neurorehabilitation exercises.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Axial completeness of chronic spinal cord injury based on spine MRI | 5 years
  Spared region volume at the injury site as assessed by spine MRI will be compared with clinical SCI score as measured by the ISCNSCI exam.
Sagittal completeness of chronic spinal cord injury based on spine MRI | 5 years
  Intramedullary lesion length will be measured via spine MRI and compared with clinical SCI score as measured by the ISCNSCI exam.
Presence of descending connections in chronic spinal cord injury based on transcranial magnetic stimulation | 5 years
  The latency of transcranial magnetic stimulation pulses will be measured via electromyography and compared with clinical SCI score as measured by the ISCNSCI exam.
Presence of ascending connections in chronic spinal cord injury based on somatosensory evoked potentials. | 5 years
  The latency of somatosensory evoked potential pulses will be measured via electromyography and compared with clinical SCI score as measured by the ISCNSCI exam.

SECONDARY OUTCOMES:
Research priorities of Veteran spinal cord injury stakeholders | 2 years
  The research priorities of Veterans with chronic spinal cord injury will be obtained and compared with previously published results in the non-Veteran population.
Voluntary motor function in the presence of non-invasive stimulation | 5 years
  Increases in electromyography will be assessed with and without the use of non-invasive transcutaneous spinal stimulation.
Sensory responses in the presence of non-invasive stimulation | 5 years
  Participants will self-report any changes in sensation during the application of non-invasive transcutaneous spinal stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Calvert, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share de-identified datasets and results collected through this proposal by depositing these data at the National Library of Medicine (NLM) PubMed Central website repository as this is a VA supported data repository. The raw and processed neurophysiological data will be shared with supplementary metadata that includes information about the study methodology used to collect the data, details about the code, and definitions of variables.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be posted following publication of the data in a scientific journal. It is anticipated that this project will produce approximately 1 publication per year after the second year, with the data published simultaneously. All of the data will be published at the conclusion of the study in five years. The deidentified data will be posted on publicly accessible servers and will be stored there permanently.
Access Criteria: Deidentified data will be accessible by all who interested parties. Any further requests will be made and reviewed by the PI.